CLINICAL TRIAL: NCT07058194
Title: Preoperative and Postoperative Erector Spinae Plane Block: Effects on Frontal QRS-T Angle in Laparoscopic Surgery - A Prospective Randomized Study
Brief Title: Effect of Pre- and Postoperative ESP Block on Frontal QRS-T Angle in Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Veli Fahri Pehlivan, Assistant Professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Veli Frontal
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cholecystectomy, Laparoscopic; Pain, Postoperative; Electrocardiography; Regional Anesthesia; Cardiac Electrophysiology
Keywords: Erector Spinae Plane Block (ESP block); Frontal QRS-T Angle; Postoperative Pain Control; Cardiac Risk; Ultrasound-guided Nerve Block; QT interval
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into three parallel groups to compare the effects of preoperative and postoperative erector spinae plane block on cardiac electrophysiological parameters.
Masking Description: This is an open-label study due to the nature of the ESP block procedure, which prevents blinding of participants and care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preoperative ESP Block Group (Experimental): Patients in this group will receive bilateral ultrasound-guided erector spinae plane (ESP) block at the T7 level with 20 mL of 0.25% bupivacaine on each side (total 40 mL) before the induction of general anesthesia. ECG will be recorded preoperatively and at 1 hour postoperatively. Frontal QRS-T angle, QT interval, QTc, Tp-e interval, and Tp-e/QTc ratio will be analyzed.
  Interventions: Procedure: Preoperative Erector Spinae Plane Block; Procedure: Standard General Anesthesia; Drug: Bupivacaine
- Postoperative ESP Block Grou (Experimental): Patients in this group will undergo standard general anesthesia. At the end of surgery, bilateral ESP block will be applied at the T7 level using 20 mL of 0.25% bupivacaine per side. ECG will be taken preoperatively and at 1 hour after surgery to evaluate changes in cardiac electrophysiologic parameters including the Frontal QRS-T angle.
  Interventions: Procedure: Postoperative Erector Spinae Plane Block; Procedure: Standard General Anesthesia; Drug: Bupivacaine
- Control Group (No ESP Block) (Active Comparator): Patients in the control group will receive standard general anesthesia only, without any regional block. Preoperative and 1-hour postoperative ECGs will be obtained for comparison of electrophysiologic markers such as Frontal QRS-T angle, QT, QTc, Tp-e, and Tp-e/QTc.
  Interventions: Procedure: Standard General Anesthesia

INTERVENTIONS:
Procedure: Preoperative Erector Spinae Plane Block — This procedure involves bilateral ultrasound-guided erector spinae plane block at the T7 level using 20 mL of 0.25% bupivacaine per side (total 40 mL) before the induction of general anesthesia. The intervention aims to evaluate the effects of preoperative ESP block on changes in frontal QRS-T angle and other ECG-derived cardiac electrophysiological parameters.
  Other Names: Bilateral ESP Block Before Induction
  Arms: Preoperative ESP Block Group
Procedure: Postoperative Erector Spinae Plane Block — Patients in this group will undergo standard general anesthesia. At the end of the surgery, bilateral ESP block will be performed under ultrasound guidance at the T7 level using 0.25% bupivacaine (20 mL per side, total 40 mL). The aim is to evaluate the effect of postoperative ESP block on changes in frontal QRS-T angle and other cardiac electrophysiological parameters.
  Other Names: Bilateral ESP Block After Surgery
  Arms: Postoperative ESP Block Grou
Procedure: Standard General Anesthesia — This group will receive standard general anesthesia without any additional regional block. ECG data will be collected preoperatively and 1 hour postoperatively to serve as a comparison for electrophysiological changes observed in the intervention groups.
  Other Names: Control
Drug: Bupivacaine — 0.25% bupivacaine, 20 mL per side (total 40 mL), administered bilaterally at T7 level under ultrasound guidance as part of ESP block.
  Other Names: used as part of ESP block interventions
  Arms: Postoperative ESP Block Grou; Preoperative ESP Block Group

SUMMARY:
This study aims to investigate the effects of preoperative and postoperative Erector Spinae Plane (ESP) block on the frontal QRS-T angle, a marker of cardiac electrophysiological instability, in patients undergoing laparoscopic cholecystectomy. A total of 120 patients aged 18-65 with ASA I-II status will be randomized into three groups: Control (no ESP), Preoperative ESP, and Postoperative ESP. Electrocardiograms (ECGs) will be obtained preoperatively and one hour postoperatively to assess changes in QRS-T angle and other repolarization parameters. This randomized controlled trial will help clarify the potential cardiac effects of ESP block depending on its timing and may provide insight into optimizing anesthetic safety in surgical patients.

DETAILED DESCRIPTION:
Erector Spinae Plane (ESP) block is widely used in laparoscopic surgeries for postoperative pain control due to its simplicity and efficacy. However, its influence on the autonomic nervous system and subsequent cardiovascular effects, including changes in cardiac electrophysiological parameters, remains insufficiently understood. The frontal QRS-T angle has emerged as a novel and reliable ECG-derived marker associated with increased cardiac risk and ventricular repolarization heterogeneity.

This prospective, randomized, controlled, single-center trial aims to evaluate the impact of ESP block timing on the frontal QRS-T angle. A total of 120 adult patients scheduled for elective laparoscopic cholecystectomy will be randomly assigned into three groups:

Control group (no ESP block),

Preoperative ESP block group,

Postoperative ESP block group.

Bilateral ESP blocks will be administered using 0.25% bupivacaine under ultrasound guidance at the T7 level. Standard general anesthesia will be applied to all patients. ECG recordings will be obtained preoperatively and at the first postoperative hour to calculate the frontal QRS-T angle, QT interval, QTc, Tp-e, Tp-e/QT, and Tp-e/QTc ratios.

The primary outcome is the change in the frontal QRS-T angle. Secondary outcomes include pain scores (VAS), analgesic consumption, and other ECG-based repolarization markers. The findings may enhance perioperative cardiac risk stratification and inform decisions on the optimal timing of ESP block administration in surgical patients with potential cardiac vulnerability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* ASA physical status I-II
* Scheduled for elective laparoscopic cholecystectomy
* Voluntary written informed consent obtained
* Normal preoperative 12-lead ECG (no conduction abnormalities or arrhythmias)

Exclusion Criteria:

* History of cardiac disease (e.g., arrhythmia, myocardial infarction, heart failure)
* Current use of medications affecting cardiac conduction (e.g., antiarrhythmics, beta-blockers)
* Known allergy to local anesthetics
* Coagulation disorders or current anticoagulant therapy
* Pregnancy or breastfeeding
* Local infection or anatomical deformity at the ESP block injection site
* Patients with psychiatric or neurological disorders impairing cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-29 (Estimated)

PRIMARY OUTCOMES:
Change in Frontal QRS-T Angle Between Preoperative and Postoperative ECG | From 1 hour before surgery to 1 hour after surgery
  The primary outcome is the change in frontal QRS-T angle measured on 12-lead ECG before surgery (baseline) and 1 hour after laparoscopic cholecystectomy. This angle is a marker of ventricular repolarization heterogeneity and potential cardiac risk.

SECONDARY OUTCOMES:
Change in QT Interval (QTc) Pre- and Postoperatively | From 1 hour before surgery to 1 hour after surgery
  The corrected QT interval (QTc) will be measured on 12-lead ECG before and 1 hour after surgery to evaluate changes in ventricular repolarization associated with ESP block.
Postoperative Pain Intensity Based on Visual Analog Scale (VAS) | At 2, 6, 12, and 24 hours postoperatively
  Pain intensity will be assessed using the 10 cm Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain), at rest and during coughing at 2, 6, 12, and 24 hours postoperatively. Higher scores indicate worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Veli F Pehlivan, Asiss Prof, Principal Investigator — Harran University Faculty of Medicine, Department of Anesthesiology
Locations (1):
- Veli Fahri Pehlivan, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study data will not be shared with other researchers. The dataset contains identifiable clinical and ECG data that are not suitable for public sharing under the current data protection regulations.